CLINICAL TRIAL: NCT06426173
Title: Effect of Resistance Training on Functional Capacity, Quality of Life and Cardiac Biomarkers in Patients on the Waiting List for Heart Transplant: a Randomized and Controlled Clinical Trial
Brief Title: Effect of Resistance Training in Patients on the Waiting List for Heart Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Rafael M. Ianotti, PT, Clinical Research Coordinator - Physiotherapy Division - Heart Institute (InCor), University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 77806024.4.0000.0068
Record Dates: First submitted 2024-04-29; First posted 2024-05-23 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Heart Transplant
Keywords: heart failure; resistance training; cardiac rehabilitation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for conducting the functional assessment will be blinded to the randomization and allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Training Group (Experimental): Patients will receive the standard treatment provided by the hospital inpatient unit alongside the resistance training program.
  Interventions: Other: Resistance Training Program; Other: Standard Treatment Group
- Standard Treatment Group (Active Comparator): Patients will receive the standard treatment provided by the hospital inpatient unit.
  Interventions: Other: Standard Treatment Group

INTERVENTIONS:
Other: Resistance Training Program — The resistance training program will be individualized and divided into four stages of increasing complexity. It will be conducted for approximately 40 minutes per day, three times a week, for 12 weeks, under supervision. Each patient will begin the program at the stage corresponding to their functional capacity. The resistance load will be set at 50% of the maximum resistance (1RM) obtained in the initial assessment. Throughout all stages of the exercise program, the target intensity will range from light (≤ 12) to moderate (≤ 15) on the Borg scale.
  Arms: Resistance Training Group
Other: Standard Treatment Group — Patients will receive the standard treatment provided by the hospital inpatient unit, which includes guidance on reducing sedentary time, encouragement to walk, and performance of active and breathing exercises when necessary.

SUMMARY:
The present longitudinal, randomized, and blinded clinical trial aims to:

* Evaluate the effects of resistance training on the functional capacity, quality of life, and cardiac biomarkers of hospitalized patients with heart failure (HF) on the waiting list for heart transplantation (HTx).
* Evaluate the associations between Fried's frailty classification and functional capacity responses to resistance training.

The protocol will have a total duration of 12 weeks.

DETAILED DESCRIPTION:
Heart failure (HF) presents a significant challenge to contemporary healthcare systems. As HF progresses, heart transplantation (HTx) becomes the primary treatment option to enhance survival rates. Patients awaiting HTx often endure extended hospitalizations and rely on continuous inotropic support. This scenario exacerbates bed rest and potentially worsening functional capacity. Resistance training has shown promise in mitigating the detrimental effects of immobility, however, limited research has explored its impact on HF patients on the HTx waiting list.

Objectives:

* To evaluate the effects of resistance training on functional capacity, quality of life, and cardiac biomarkers in hospitalized patients with HF on the HTx waiting list.
* To assess the associations between Fried's frailty phenotype and functional capacity responses to resistance training, hemodynamic behavior during the protocol, and the incidence of adverse events during the protocol implementation.

Methods:

A total of 50 patients hospitalized on the HTx waiting list will be recruited for this study. Participants will be randomly assigned to one of two groups: the resistance training group (TG) and the control group (CG). Assessments will occur at three time points: baseline (T0), at 6 weeks (T1), and at 12 weeks (T2) of resistance training. Clinical parameters will be evaluated, including the six-minute walk test and the Short Physical Performance Battery. Peripheral muscle strength will be measured using a dynamometer, and inspiratory muscle strength will be assessed through maximum inspiratory pressure. Quality of life will be evaluated using the Kansas City Cardiomyopathy Questionnaire-12. Additionally, cardiac biomarkers, such as exhaled air ketone and brain natriuretic peptide levels in venous blood samples, will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients included in heart transplant list ≤1 month
* hemodynamically stable in the last 48 hours defined as mean arterial pressure (MAP) ≥ 60 mmHg and ≤ 120 mmHg and - Heart rate (HR) ≥ 60 bpm and ≤ 120 mmHg.
* dobutamine dose ≤ 10 mcg/kg/min

Exclusion Criteria:

* heart failure of arrhythmogenic and/or restrictive etiology
* presence of uncontrolled acute arrhythmias
* cognitive, orthopedic, or neuromotor changes that prevent functional tests from being carried out

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To investigate changes in physical performance measured by Six-Minute Walk Test. | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Measures: the assessment will take place in a flat 30-meter corridor, marked every 1 meter with non-slip flooring, and the patient will be instructed to walk for six minutes as fast as possible.
To investigate changes in physical performance measured by Short Physical Performance Battery (SPPB). | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  The SPPB consists of three additional tests assessing balance, mobility, and strength. Each test is scored from 0 (indicating a worse outcome) to 4 (indicating a better outcome) points. At the completion of all tests, the total score ranges from 0 to 12 points.
To investigate changes in respiratory muscle strength: | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Maximum inspiratory pressure (measured in cmH2O)
To investigate changes in peripheral muscle strength. | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Handgrip test (measured in KgF)
To investigate changes in quality of life: | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Kansas City Cardiomyopathy Questionnaire-Short Version. The total score ranges from 0 (indicating a worse outcome) to 100 (indicating a better outcome) points.
Enhancing the investigation of changes in cardiac biomarker ketones | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Ketones in exhaled air (measured in μg/L)
Enhancing the investigation of changes in cardiac biomarker brain natriuretic peptide | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  Brain natriuretic peptide in venous blood sample (picogram per milliliter, pg/ml)

SECONDARY OUTCOMES:
To investigate changes Fried's frailty phenotype | The data will be collected on the baseline (T0), at 6 weeks (T1), and at 12 weeks (T2).
  The Fried's frailty phenotype scale ranges from 0 to 5 points, where: 0 points denote non-frailty, up to 2 points denote pre-frailty, and ≥3 points denote frailty
To investigate changes in heart rate( bpm) | Immediately before and after each session exercise training.(3 times per week, during 12 weeks)
To investigate changes in blood pressure (mmHg) | Immediately before and after each session exercise training (3 times per week, during 12 weeks)
To investigate changes in perceived exertion sensation: | Immediately before and after each session exercise training.(3 times per week, during 12 weeks)
  Borg Rating of Perceived Exertion (0-lower, up to 10- highest)
To investigate the occurrence of adverse events:Hemodynamic instability | In each intervention period (3 days a week for 12 weeks)
  Hemodynamic instability ( MAP < 60 mmHg or >120 mmHg)
To investigate the occurrence of adverse events:Arrhythmia | In each intervention period (3 times per week for 12 weeks)
  Heart rate ( HR < 50 bpm or > 120 bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Juliana A Nascimento, PT, PhD, Principal Investigator — University of Sao Paulo; Rafael M Ianotti, PT, Principal Investigator — Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil